CLINICAL TRIAL: NCT05462535
Title: An Observational Study to Evaluate the Efficacy and Safety of Amosartan Plus Tablet in Uncontrolled Essential Hypertension Patients
Brief Title: An Observational Study to Evaluate Effectiveness and Safety of Amosartan Plus Tablet
Status: Completed | Type: Observational
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: HM-AMOP-OS-01
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Hypertension,Essential
MeSH Terms: conditions — Essential Hypertension | interventions — Tablets; Losartan; Chlorthalidone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm, Single group(No interventional): Observational
  Interventions: Drug: Amosartan Plus Tab.

INTERVENTIONS:
Drug: Amosartan Plus Tab. — Amosartan Plus Tab., Once daily administered per the locally approved product information
  Other Names: Amlodipine camsylate, Losartan potassium, Chlorthalidone

SUMMARY:
This study was to evaluate the therapeutic effect and safety of Amosartan Plus tablet administration in uncontrolled essential hypertension patients.

During the routine medical visit, Amosartan Plus tablets were administered to patients in need of blood pressure control according to the investigator's judgment.

In this study, effectiveness and safety information of treatment of Amosartan Plus tablets was followed for 6 months (up to 12 months), and observation of the target patients was terminated after collecting relevant data.

As this study was a non-interventional observational study, all patients received prescriptions according to the routine treatment procedure, and there were no visits or procedures required according to the observational study protocol.

DETAILED DESCRIPTION:
This study was a multi-center, prospective, non-interventional, observational study of factors affecting blood pressure after treatment with Amosartan Plus tablet in uncontrolled essential hypertension patients.

Data was collected from patients receiving routine treatment at hospitals in South Korea. Each patient visited the institution according to the protocol that designed the follow-up visits for six months to examine the effectiveness and safety of Amosartan Plus tablet.

This study approved by the institutions' IRBs and was conducted in compliance with clinical research ethics regulations.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled essential hypertension patients
* Those who have already decided to administer Amosartan Plus tablet under the medical judgment of the researcher
* Those who voluntarily decided to participate in this study and consented in writing to the consent form

Exclusion Criteria:

* Patients for whom use of Amosartan Plus tablet is prohibited

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Uncontrolled essential hypertension patients
Sampling Method: Non-Probability Sample
Enrollment: 4785 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in SBP/DBP | 24 weeks
Percentage from baseline in SBP/DBP | 24 weeks
Percentage of patients achieving target blood pressure | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi Pharmaceutical Company Limited, Seoul, South Korea